CLINICAL TRIAL: NCT01988415
Title: A Prospective Study to Evaluate the Feasibility of a New Treatment Algorithm for Wavefront-Guided Lasik Correction of Myopic Refractive Errors
Brief Title: New Treatment Algorithm to Reduce Spherical Aberration After LASIK Correction for Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STAR-114-SARA
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- VSS-Rx1 OPM vs Commercial iDesign Treatment (Other): Commercially available iDesign treatment planning software used to calculate the LASIK treatment profile in one eye (active comparator [i.e., control]) and investigational software (includes a modified algorithm designed to reduce the induction of postoperative spherical aberration) in the fellow eye (experimental).
  Interventions: Device: VSS-Rx1 OPM vs Commercial iDesign Treatment

INTERVENTIONS:
Device: VSS-Rx1 OPM vs Commercial iDesign Treatment — Commercially available iDesign treatment planning software used to calculate the LASIK treatment profile vs VSS-Rx1 OPM (includes a modified algorithm designed to reduce the induction of postoperative spherical aberration).

SUMMARY:
The purpose of this clinical trial is to demonstrate that treatments generated by an investigational algorithm reduces spherical aberration compared to currently available iDesign treatments.

DETAILED DESCRIPTION:
Post-LASIK induction of spherical aberration is currently among the most prominent challenges for refractive surgery. The presence of significant spherical aberration in the visual system results in reduced contrast sensitivity, visual symptoms such as "glare" and "halos," and "night myopia" or the induction of myopia under low lighting (larger pupil size). A modified Treatment Planning Software (TPS) "VSS-Rx1 OPM software" has been developed that uses a modified algorithm (software that designs the LASIK treatment profile) to limit the induction of postoperative spherical aberration. Commercially available software used to calculate the LASIK treatment profile was used in one eye (active comparator [i.e., control]) and VSS-Rx1 OPM software was used in the fellow eye (experimental). Subjects were masked to the use of either the commercially available or VSS-Rx1 OPM software.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at the time of preoperative exam
* Best Spectacle Corrected Visual Acuity (BSCVA) of 20/20 or better
* Demonstration of refractive stability
* Anticipated postoperative stromal bed thickness of at least 250 microns
* Willing and able to return for all study examinations

Exclusion Criteria:

* Pregnant, breast-feeding, or intend to become pregnant over the course of the study
* Concurrent use of topical or systemic medications that may impair healing
* History of prior intraocular or corneal surgery, active ophthalmic disease, or other ocular abnormality
* Evidence of keratoconus, corneal irregularity, or abnormal topography in the operative eye(s)
* Known sensitivity or inappropriate responsiveness to any of the medications used in the postoperative course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Tamayo, M.D., Principal Investigator — Medico Oftalmologo
Locations (1):
- Gustavo Tamayo, M.D., Bogota Laser, Bogota, Colombia

RESULTS

PARTICIPANT FLOW:
Groups:
- VSS-Rx1 OPM vs Commercial iDesign Treatment: Commercially available software used to calculate the LASIK treatment profile in one eye (active comparator [i.e., control]) and investigational software (includes a modified algorithm designed to reduce the induction of postoperative spherical aberration) in the fellow eye (experimental).
Period: Overall Study
Arm/Group | VSS-Rx1 OPM vs Commercial iDesign Treatment
Started | 26 (52 eyes of 26 subjects (paired-eyes: commercial and investigational software))
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This was a paired-eye study in which treatment of 26 participants included both eyes (52 eyes total). Use of the commercial versus VSS-Rx1 OPM treatment planning software was randomized by eye. One eye of each subject received the investigational treatment and the fellow eye received the commercial treatment.
Arm/Group | VSS-Rx1 OPM vs Commercial iDesign Treatment
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Region of Enrollment [Number; unit: participants]
  Colombia | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Postoperative Spherical Aberration
Description: Primary Efficacy Outcome Measure: mean spherical aberration of eyes treated with the VSS-Rx1 OPM treatment planning software compared to that of eyes treated with the commercial iDesign treatment planning software.
Time Frame: 3 months
Population: The analysis population was all evaluable eyes.
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Groups:
- Commercial iDesign Treatment Planning Software: Commercial iDesign treatment planning software: perform wavefront-guided LASIK based upon measurements obtained with the iDesign System and the commercial iDesign treatment planning software
- VSS-Rx1 OPM Treatment Planning Software: Investigational treatment planning software: perform wavefront-guided LASIK based upon measurements obtained with the iDesign System and the VSS-Rx1 OPM treatment planning software
Arm/Group | Commercial iDesign Treatment Planning Software | VSS-Rx1 OPM Treatment Planning Software
Number analyzed (Participants) | 26 | 26
Number analyzed (Eyes) | 26 | 26
µm | 0.069 (0.092) | 0.016 (0.108)

2. Primary Outcome: Percentage of Eyes Losing More Than 2 Lines of Best-corrected Distance Visual Acuity
Description: Primary Safety Outcome Measure: percentage of eyes losing more than 2 lines of best-corrected distance visual acuity
Time Frame: 3 Months
Population: The analysis population was all evaluable eyes.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Commercial iDesign Treatment Planning Software | VSS-Rx1 OPM Treatment Planning Software
Number analyzed (Participants) | 26 | 26
Number analyzed (Eyes) | 26 | 26
percentage of eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Commercial iDesign Treatment Planning Software | VSS-Rx1 OPM Treatment Planning Software
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall have the first right of publication of study data for the first 12 months. The institution or principal investigator may not disclose any of the Sponsor's proprietary information.